CLINICAL TRIAL: NCT01770847
Title: Diurnal Variations in Arterial Stiffness in Patients With Chronic Kidney Disease and Healthy Age Matched Controls
Brief Title: Arterial Stiffness in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 12\SS\0088
Record Dates: First submitted 2012-11-28; First posted 2013-01-18 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy controls: Healthy age matched controls
- Chronic kidney diease: Chronic kidney disease patients stage 2-4

SUMMARY:
Diurnal variations in the cardiovascular system apparent in healthy individuals, are different in chronic kidney disease patients. Therefore, diurnal variations in arterial stiffness may also differ in chronic kidney disease patients. This study aims to identify and evaluate diurnal variations in arterial stiffness in chronic kidney disease patients and compare them to those in age matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure <160 whether or not on antihypertensive medication
* diastolic blood pressure <100mmHg whether or not on antihypertensive medication
* Chronic kidney disease stage 2-5

Exclusion Criteria:

* Systolic blood pressure ≥160mmHg
* Diastolic blood pressure ≥100mmhg
* Significant comorbidity (investigator opinion but to include alcoholism and terminal illness)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential patients will be identified from renal clinics at the Royal Infirmary and Western General Hospital. Suitable participants will initially be identified by a member of the direct healthcare team.
  Healthy volunteers will be indentified through the Clinical Research Centre community database and poster advertising at the University of Edinburgh.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Diurnal variations in arterial stiffness | Over one 26 hour period arterial stiffness measurements will be obtained every 30 minutes from 7am to 12am and every 60 minutes from 12am to 7am
  The principal objective of this study is to evaluate whether diurnal variations in arterial stiffness are blunted in chronic kidney disease compared to healthy age matched controls

SECONDARY OUTCOMES:
Diurnal variations in aortic and brachial blood pressure | Over one 26 hour period blood pressure measurements will be obtained every 30 minutes from 7am to 12am and every 60 minutes from 12am to 7am
  Secondary objective of this study is to evaluate whether diurnal variations in aortic and brachial blood pressure are blunted in chronic kidney disease compared to healthy age matched controls
Relationship between changes in blood pressure and arterial stiffness | Over one 26 hour period
  Secondary objective of this study is to evaluate whether diurnal variations in arterial stiffness are dependent on changes in blood pressure in both chronic kidney disease patients and age matched controls.

CONTACTS AND LOCATIONS:
Overall Officials: David J Webb, MB BS MD DSc FRCP FRSE FMedSci, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical Research Centre, 2nd Floor Western General Hospital, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Dhaun N, Moorhouse R, MacIntyre IM, Melville V, Oosthuyzen W, Kimmitt RA, Brown KE, Kennedy ED, Goddard J, Webb DJ. Diurnal variation in blood pressure and arterial stiffness in chronic kidney disease: the role of endothelin-1. Hypertension. 2014 Aug;64(2):296-304. doi: 10.1161/HYPERTENSIONAHA.114.03533. PMID 24890823